CLINICAL TRIAL: NCT05245214
Title: Comprehensive Analysis Of Muscle Wasting In Disc Herniation
Brief Title: Muscle Analyze In Patient With Disc Herniation
Status: Completed | Type: Observational
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Ayşenur Gökşen, Assistant Prof, Karamanoğlu Mehmetbey University
Other Study IDs: 06-2021/30
Record Dates: First submitted 2022-01-10; First posted 2022-02-17 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Disk Herniated Lumbar
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with disc herniation: Having only disc degeneration and not having any other neurological or orthopedic disease. Patients who had previous spinal surgery, patients with lumbar scoliosis, spondylolisthesis or structural defect in the sacrum were excluded from the study.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging
- Patient in control group: Patients without disc herniation, severe disc degeneration and spondylolisthesis were included in the control group.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — Muscle analysis by Magnetic Resonance Imaging

SUMMARY:
This study which was planned to investigate the factors affecting m. erector spinae (ES), m. multifidus (MF), m. psoas major (PM) and m. quadratus lumborum (QL), which stabilize the lumbar region in the case of disc herniation. In this study, the effects of disc herniation, herniation severity, age, and spinal biomechanics were investigated.

DETAILED DESCRIPTION:
This study was carried out on 330 individuals with and without lumbar disc herniation. All individuals were divided into 3 groups according to their age. The inclusion criteria: Having only disc degeneration and not having any other neurological or orthopedic disease. Patients who had previous spinal surgery, patients with lumbar scoliosis, spondylolisthesis or structural defect in the sacrum were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Having only disc degeneration and not having any other neurological or orthopedic disease. Patients who had previous spinal surgery, patients with lumbar scoliosis, spondylolisthesis or structural defect in the sacrum were excluded from the study.

Exclusion Criteria:

* Patients who had previous spinal surgery, patients with lumbar scoliosis, spondylolisthesis or structural defect in the sacrum were excluded from the study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients without disc herniation, severe disc degeneration and spondylolisthesis were also withdrawn from the System and included in the control group. 80 individuals with aged between 20-70 years included control group.
Sampling Method: Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Muscle cross-area | 1 Month
  The cross-sectional area of the Multifidus, Erector Spina, Quadratus Lumborum, and Psoas Major muscles on both sides were measured using the T2-weighted axial Magnetig Resonance Imaging.

SECONDARY OUTCOMES:
Lumbar Biomechanic | 1 Month
  Biomechanic analysis was performed by measuring the sagittal curve using T2-weighted sagittal images.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Gökşen, PhD, Principal Investigator — Karamanoğlu Mehmetbey University
Locations (1):
- Karamanoğlu Mehmetbey University, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study was planned to investigate the factors affecting muscle which stabilize the lumbar region in the case of disc herniation.

REFERENCES:
- [Background] Sun D, Liu P, Cheng J, Ma Z, Liu J, Qin T. Correlation between intervertebral disc degeneration, paraspinal muscle atrophy, and lumbar facet joints degeneration in patients with lumbar disc herniation. BMC Musculoskelet Disord. 2017 Apr 20;18(1):167. doi: 10.1186/s12891-017-1522-4. PMID 28427393